CLINICAL TRIAL: NCT00283062
Title: A Multicenter, Open-Label, Randomized, Phase III Trial Comparing Immediate Adjuvant Hormonal Therapy (ELIGARD®- Leuprolide Acetate) in Combination With TAXOTERE® (Docetaxel) Administered Every Three Weeks Versus Hormonal Therapy Alone Versus Deferred Therapy Followed by the Same Therapeutic Options in Patients With Prostate Cancer at High Risk of Relapse After Radical Prostatectomy
Brief Title: Adjuvant Leuprolide With or Without Docetaxel in High Risk Prostate Cancer After Radical Prostatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976J_3501; EudraCT # : 2004-002203-32; NCT00343967 (obsolete NCT alias)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2010-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Drug Therapy; Leuprolide; luprolide acetate gel depot

ARMS (4):
- Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) (Experimental): Participants administered docetaxel every three weeks (q3w) for 6 cycles in combination with leuprolide acetate every 3 months for 18 months immediately following prostatectomy.
  Interventions: Drug: Docetaxel (TAXOTERE®) Chemotherapy; Drug: Leuprolide acetate ( ELIGARD®) Hormonal Therapy
- Leuprolide Acetate - Immediate Treatment (I-HT) (Active Comparator): Participants administered leuprolide acetate every 3 months for 18 months immediately following prostatectomy.
  Interventions: Drug: Leuprolide acetate ( ELIGARD®) Hormonal Therapy
- Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) (Experimental): Participants in whom treatment was deferred from randomization until first progression - i.e. PSA progression and/or radiologically or histologically documented progression. Participants were treated with docetaxel every three weeks (q3w) for 6 cycles in combination with leuprolide acetate every 3 months for 18 months.
  Interventions: Drug: Docetaxel (TAXOTERE®) Chemotherapy; Drug: Leuprolide acetate ( ELIGARD®) Hormonal Therapy
- Leuprolide Acetate - Deferred Treatment (D-HT) (Active Comparator): Participants in whom treatment was deferred from randomization until first progression - i.e. PSA progression and/or radiologically or histologically documented progression. Participants were treated with with leuprolide acetate every 3 months for 18 months.
  Interventions: Drug: Leuprolide acetate ( ELIGARD®) Hormonal Therapy

INTERVENTIONS:
Drug: Docetaxel (TAXOTERE®) Chemotherapy — 75 mg/m^2 docetaxel administered intravenously over 1 hour on Day 1 every three weeks (q3w) for 6 cycles. The first cycle was to be administered within 8 days after randomization.
  Corticosteroid pre-medication was mandatory. The following schedule was recommended - 8 mg Dexamethasone orally for 6 doses given - the night before chemotherapy, the morning of chemotherapy, 1 hour before docetaxel infusion, the night of chemotherapy, the morning of the day after chemotherapy and the night of the day after chemotherapy.
  Arms: Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT)
Drug: Leuprolide acetate ( ELIGARD®) Hormonal Therapy — 22.5 mg leuprolide acetate injection administered subcutaneously (SC) every 3 months for 18 months. The first injection was to be administered within 8 days after randomization.
  Arms: Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT); Leuprolide Acetate - Immediate Treatment (I-HT)
Drug: Docetaxel (TAXOTERE®) Chemotherapy — 75 mg/m^2 docetaxel administered IV over 1 hour on Day 1 q3w for 6 cycles. The first cycle was to be administered within 30 days after progression was confirmed.
  Corticosteroid pre-medication was mandatory. The following schedule was recommended - 8 mg Dexamethasone orally for 6 doses given - the night before chemotherapy, the morning of chemotherapy, 1 hour before docetaxel infusion, the night of chemotherapy, the morning of the day after chemotherapy and the night of the day after chemotherapy.
  Arms: Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT)
Drug: Leuprolide acetate ( ELIGARD®) Hormonal Therapy — 22.5 mg leuprolide acetate injection administered subcutaneously (SC) every 3 months for 18 months. The first injection was to be administered within 30 days after progression is confirmed (on Day 1 of docetaxel administration).
  Arms: Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT)
Drug: Leuprolide acetate ( ELIGARD®) Hormonal Therapy — 22.5 mg leuprolide acetate injection administered subcutaneously (SC) every 3 months for 18 months. The first injection was to be administered within 30 days after progression is confirmed.
  Arms: Leuprolide Acetate - Deferred Treatment (D-HT)

SUMMARY:
This is a prospective, multicenter, open-label, randomized phase III study in participants at high risk of recurrent prostate cancer after radical prostatectomy. The study will investigate

* Treatment with docetaxel (TAXOTERE®) every three weeks (q3w) plus leuprolide acetate (ELIGARD®) versus leuprolide acetate alone (ELIGARD®)
* Immediate treatment following prostatectomy versus deferred treatment at the time of relapse

Using a 2x2 factorial design participants will therefore be randomized to

* Immediate adjuvant treatment with docetaxel plus leuprolide acetate (chemotherapy and hormonal therapy)
* Immediate adjuvant treatment with leuprolide acetate alone (hormonal therapy)
* Deferred treatment with docetaxel plus leuprolide acetate (chemotherapy and hormonal therapy)
* Deferred treatment with leuprolide acetate alone (hormonal therapy)

Primary Objective:

* The primary objective of the study is to compare progression-free survival using a 2x2 factorial design

Secondary Objectives:

* To compare the 5-year overall, cancer-specific and metastasis-free survival after systemic treatment between the groups
* To compare the safety and tolerability between Docetaxel in combination with leuprolide acetate and leuprolide acetate alone.
* To evaluate quality of life as measured by the FACT-P questionnaire.

Originally, 1696 participants were planned in the study (with 424 participants randomized to each arm). However, only a total of 211 participants completed the randomization procedure as of 26 September 2007. Thus, sanofi-aventis, in accordance with the Steering Committee, decided to stop the participant recruitment as of 26 September 2007. Participants who had already signed their Informed Consent (IC) before September 26, 2007 were allowed to enter the randomization if they met eligibility criteria. The final revised number of planned participants to be randomly assigned to the 4 treatment arms was 250, and 228 participants were actually randomized.

The final sample size did not allow all the statistical analyses to be conducted on efficacy data. Therefore, the protocol was amended to reflect the change in the plans for statistical analysis. The study was underpowered to serve as the basis for drawing conclusions regarding efficacy and quality of life (QoL) endpoints.

DETAILED DESCRIPTION:
The study consisted of the following:

* Randomization of eligible participants within 120 days of prostatectomy
* For participants assigned to immediate therapy, a treatment period up to 18 months within 8 days of randomization
* For participants assigned to deferred treatment, a treatment period up to 18 months after evidence of progression prior to December 2010. Participants who did not progress before December 2010 were withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

Participants who met all of the following criteria were considered for enrollment into the study.

* Pathologically confirmed adenocarcinoma of the prostate based on central pathology review. All other variants are excluded
* Randomization should occur less than 120 days after prostatectomy AND lymphadenectomy.
* A predicted probability of 5-year freedom from progression ≤ 60%, as determined by the postoperative nomogram developed by M. Kattan.
* Bone-scan without evidence of metastasis (within 6 months of randomization)
* Chest x-ray without evidence of metastasis (within 6 months of randomization)
* Abdominal computed tomography (CT) Scan without evidence of metastasis (within 6 months of randomization)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Hematology evaluation within 2 weeks prior to randomization:

  * Neutrophils ≥ 2,000/mm3
  * Hemoglobin ≥ 10 g/dL
  * Platelets ≥ 100,000/mm3
* Hepatic and renal function evaluation within 2 weeks prior to randomization:

  * Serum creatinine ≤1.5 × Upper normal limit (UNL) for the institution. If serum creatinine is > 1.5 × UNL, calculate creatinine clearance (should be ≥ 60ml/minute).
  * Total serum bilirubin ≤ UNL for the institution. Participants with Gilbert's syndrome may be eligible if indirect serum bilirubin levels at the time of randomization and, at least 6 month prior to randomization, confirm this condition (i.e. elevated indirect serum bilirubin).
  * Serum glutamic oxaloacetic transaminase (SGOT) and/or serum glutamic pyruvic transaminase (SGPT) ≤ 1.5 × institutional UNL if alkaline phosphatase is ≤ UNL OR
  * alkaline phosphatase ≤ 5 × UNL if SGOT and SGPT are ≤ UNL
* Prostate Specific Antigen (PSA) evaluation within 9 months prior to prostatectomy. However, a 120-day timeframe is recommended
* Post operative PSA necessary for eligibility is defined as a level ≤ 0.2ng/mL using a standard assay at least 30 days after radical prostatectomy and within 7 days prior to randomization. Note that randomization should occur within 120 days after radical prostatectomy
* Serum testosterone ≥ 150ng/dL within 6 months prior to randomization.

Exclusion Criteria:

Participants presenting with any of the following will not be included in the study.

* Prior systemic treatment for prostate cancer with hormonal therapy, chemotherapy, or any other anticancer therapy.
* Prior radiation therapy.
* Participants who received, are receiving or scheduled to receive post-operative radiotherapy.
* Participants taking alternative therapies for cancer must stop taking these therapies prior to randomization. Alternative therapies are not allowed during the treatment or follow-up portions of the study. This includes (but is not limited to) alternative therapies such as :

  * PC-SPES (all types)
  * 5-alpha reductase inhibitors
* Bisphosphonates are to be stopped prior to randomization and are not allowed during the study.
* Chronic treatment with corticosteroids unless initiated > 6 months prior to study entry and at low dose ( ≤ 20 mg methylprednisolone per day or equivalent).
* History of a malignancy other than prostate cancer. Exceptions to these criteria include:

  * participants with adequately treated non-melanoma skin cancers, and
  * participants with a history of another malignancy that was curatively treated (including participants with superficial bladder cancer) and who have not had evidence of disease for a minimum of 5 years.
* Peripheral neuropathy ≥ Grade 2.
* Electrocardiogram (ECG) with significant abnormalities (as determined by the investigator) within 90 days prior to randomization.
* Participants who are medically unstable, including but not limited to active infection, acute hepatitis, gastrointestinal bleeding, uncontrolled cardiac arrhythmias, interstitial lung disease, inflammatory bowel disease, uncontrolled angina, uncontrolled hypercalcemia, uncompensated congestive heart failure, uncontrolled diabetes, dementia, seizures, superior vena cava syndrome.
* Participants with history of hypersensitivity to polysorbate 80.
* Participants with a known history of viral hepatitis (B, C).

The above information was not intended to contain all considerations relevant to potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Aussel, Study Director — Sanofi
Locations (17):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Québec, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico
- Sanofi-Aventis Administrative Office, PE Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Gauteng, South Africa
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Originally, the study was planned for 1696 participants to be randomized. However, enrollment was not met and in September 2007, the Steering Committee decided to stop recruitment. Only participants who had signed Informed Consent by then and met eligibility criteria were randomized. 228 participants were randomized to this study.
Groups:
- Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT): Participants administered 75 mg/m^2 docetaxel every three weeks (q3w) for 6 cycles in combination with 22.5 mg leuprolide acetate every 3 months for 18 months immediately following prostatectomy.
- Leuprolide Acetate - Immediate Treatment (I-HT): Participants administered 22.5 mg leuprolide acetate every 3 months for 18 months immediately following prostatectomy.
- Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT): Participants in whom treatment was deferred from randomization until first progression - i.e. PSA progression and/or radiologically or histologically documented progression. Participants were treated with 75 mg/m^2 docetaxel every three weeks (q3w) for 6 cycles in combination with 22.5 mg leuprolide acetate every 3 months for 18 months.
- Leuprolide Acetate - Deferred Treatment (D-HT): Participants in whom treatment was deferred from randomization until first progression - i.e. PSA progression and/or radiologically or histologically documented progression. Participants were treated with 22.5 mg leuprolide acetate every 3 months for 18 months.
Period: Overall Study
Arm/Group | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) | Leuprolide Acetate - Immediate Treatment (I-HT) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) | Leuprolide Acetate - Deferred Treatment (D-HT)
Started | 55 | 55 | 56 | 62
ADMINISTERED STUDY TREATMENT | 50 | 51 | 20 | 17
COMPLETED HORMONAL THERAPY (6 Cycles) | 44 | 48 | 15 | 13
COMPLETED CHEMOTHERAPY (6 Cycles) | 43 | 0 (Not applicable, since participants in this arm did not receive chemotherapy.) | 15 | 0 (Not applicable, since participants in this arm did not receive chemotherapy.)
Completed | 43 | 48 | 15 | 13
Not Completed | 12 | 7 | 41 | 49
Not completed — Did not receive any study medication | 5 | 4 | 36 | 45
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Progressive disease | 0 | 0 | 1 | 0
Not completed — Participant did not wish to continue | 3 | 2 | 1 | 0
Not completed — Undefined | 0 | 1 | 1 | 4
Not completed — chemotherapy not completed (cycle 6) | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) | Leuprolide Acetate - Immediate Treatment (I-HT) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) | Leuprolide Acetate - Deferred Treatment (D-HT) | Total
Number analyzed (Participants) | 55 | 55 | 56 | 62 | 228
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (7.4) | 61.6 (7.0) | 62.1 (7) | 62.9 (7.5) | 61.9 (7.2)
Age, Customized [Number; unit: participants]
  <65 years | 37 | 34 | 35 | 35 | 141
  >=65 years | 18 | 21 | 21 | 27 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 55 | 55 | 56 | 62 | 228
Race/Ethnicity, Customized [Number; unit: participants]
  White | 48 | 49 | 43 | 59 | 199
  Black | 6 | 3 | 7 | 2 | 18
  Asian/Oriental | 0 | 1 | 4 | 0 | 5
  Multiracial | 0 | 0 | 2 | 0 | 2
  Other | 1 | 2 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Assessment - Number of Participants With Disease Progression
Description: PFS is the interval from the date of surgery to date of progression. The date of progression was the earlier of
  * first PSA increase to ≥ 0.4 ng/mL confirmed within two weeks
  * date of the nadir, if PSA nadir did not reach < 0.4 ng/mL (for deferred arm)
  * first radiological/ histological evidence of tumor progression
  * death. Median PFS was to be estimated using Kaplan-Meier curves. However, enrollment was not met, and meaningful conclusions for efficacy or QoL could not be drawn. Median PFS could not be estimated. Reported is the number of participants with disease progression.
Time Frame: from the date of surgery up to 3 years after randomization of the last participant
Population: Intent-to-treat (ITT) population: all randomized participants, regardless of whether or not they received any study drug.
Measure: Number; unit: participants
Arm/Group | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) | Leuprolide Acetate - Immediate Treatment (I-HT) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) | Leuprolide Acetate - Deferred Treatment (D-HT)
Number analyzed (Participants) | 55 | 55 | 56 | 62
participants | 10 | 14 | 9 | 8

2. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival (OS) was the time interval from the date of surgery to the date of death due to any cause.
  Median OS was to be estimated using Kaplan-Meier Curves. However, enrollment was not met, and meaningful conclusions for efficacy or QoL could not be drawn. Moreover, median OS could not be estimated. Reported is the number of participants who died from any cause.
Time Frame: from the date of surgery up to 3 years after randomization of the last participant
Population: Intent-to-treat (ITT) population: all randomized participants, regardless of whether or not they received any drug.
Measure: Number; unit: participants
Arm/Group | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) | Leuprolide Acetate - Immediate Treatment (I-HT) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) | Leuprolide Acetate - Deferred Treatment (D-HT)
Number analyzed (Participants) | 55 | 55 | 56 | 62
participants | 0 | 2 | 1 | 1

3. Secondary Outcome: Median Cancer-specific Survival (CSS)
Description: The CSS was the time from the date of surgery to the date of death due to prostate cancer.
  Median CSS was to be estimated using Kaplan-Meier curves. However, enrollment was not met, and meaningful conclusions for efficacy or QoL could not be drawn. Therefore, based on a protocol amendment, median CSS was not estimated.
Time Frame: from the date of surgery up to 3 years after randomization of the last participant
Population: Based on a protocol amendment, analysis for Median CSS was not to be performed as the study was underpowered.
Measure: Number; unit: participants
Arm/Group | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) | Leuprolide Acetate - Immediate Treatment (I-HT) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) | Leuprolide Acetate - Deferred Treatment (D-HT)
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Median Metastasis-free Survival (MFS)
Description: MFS was the interval from the date of surgery to the date of the first clinical evidence of metastasis after treatment initiation. Metastasis was evaluated by a physical exam or radiologically on bone scan or CT scan. Local (palpable) progression, documented histologically or by imaging techniques was considered evidence of progression.
  Median MFS was to be estimated using Kaplan-Meier curves. However, enrollment was not met, and meaningful conclusions for efficacy or QoL could not be drawn. Therefore, based on a protocol amendment, median MFS was not estimated.
Time Frame: from the date of surgery up to 3 years after randomization of the last participant
Population: Based on a protocol amendment, analysis for Median MFS was not to be performed as the study was underpowered.
Measure: Number; unit: participants
Arm/Group | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) | Leuprolide Acetate - Immediate Treatment (I-HT) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) | Leuprolide Acetate - Deferred Treatment (D-HT)
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: To Evaluate Quality of Life (QoL) as Measured Using a Functional Assessment of Cancer Therapy-Prostate (FACT-P) Questionnaire
Description: The FACT-P is a 39-item participant questionnaire which assesses physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and additional prostate cancer specific concerns (12 items). All items are scored from 0 (not at all) to 4 (very much). The total FACT-P score ranges from 0-156, with higher scores representing a better QoL with fewer symptoms. A score of 156 represents the best outcome.
  Note: Enrollment was not met, and meaningful conclusions for efficacy or QoL could not be drawn due to the low sample size.
Time Frame: from 30 days before randomization (baseline) and 18 months after treatment initiation (for change from baseline)
Population: QoL population: The subset of randomized participants who had an evaluable baseline questionnaire and at least one evaluable post-baseline questionnaire. A baseline QoL questionnaire was considered evaluable if it was filled out within 30 days prior to randomization, and no later than the date of randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) | Leuprolide Acetate - Immediate Treatment (I-HT) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) | Leuprolide Acetate - Deferred Treatment (D-HT)
Number analyzed (Participants) | 40 | 48 | 15 | 15
score on a scale
  Baseline | 124.0 (6.0) | 121.5 (17.8) | 114.7 (13.9) | 119.7 (15.8)
  Change from Baseline (N=33, N=41, N=12, N=10) | 0.7 (12.6) | 1.7 (17.2) | 6.7 (15.9) | 6.1 (18.9)

6. Secondary Outcome: Assessment of Safety and Tolerability - Number of Participants With Adverse Events (AE)
Description: Number of participants with treatment-emergent adverse events (TEAE). A TEAE was as any adverse event that occurred or worsened during the on-treatment period, which was the period from the day of first infusion of study treatment until 30 days after the last infusion of study treatment.
Time Frame: from treatment initiation up to 19 months after treatment initiation
Population: Safety population: all randomized participants who received any study drug
Measure: Number; unit: participants
Arm/Group | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) | Leuprolide Acetate - Immediate Treatment (I-HT) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) | Leuprolide Acetate - Deferred Treatment (D-HT)
Number analyzed (Participants) | 50 | 51 | 20 | 17
participants
  with any adverse event (AE) | 47 | 48 | 19 | 14
  with any serious adverse event (SAE) | 12 | 8 | 5 | 2
  with an SAE resulting in death | 0 | 0 | 0 | 0
  with a drug-related AE | 47 | 43 | 18 | 10
  with a drug-related SAE | 6 | 0 | 2 | 0
  with AE leading to discontinue all study therapy | 2 | 0 | 1 | 0
  with AE leading to chemotherapy discontinuation | 1 | NA — Did not receive chemotherapy | 1 | NA — Did not receive chemotherapy
  with AE leading to chemotherapy dose reduction | 5 | NA — Did not receive chemotherapy | 2 | NA — Did not receive chemotherapy

ADVERSE EVENTS:
Arm/Group | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) | Leuprolide Acetate - Immediate Treatment (I-HT) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) | Leuprolide Acetate - Deferred Treatment (D-HT)
Serious Adverse Events (participants affected / at risk) | 12/50 | 8/51 | 5/20 | 2/17
Other Adverse Events (participants affected / at risk) | 47/50 | 48/51 | 19/20 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) (N=50) | Leuprolide Acetate - Immediate Treatment (I-HT) (N=51) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) (N=20) | Leuprolide Acetate - Deferred Treatment (D-HT) (N=17)
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Extravasation (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0
Optic neuropathy (Eye disorders) | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1
Respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel / Leuprolide Acetate - Immediate Treatment (I-CHT) (N=50) | Leuprolide Acetate - Immediate Treatment (I-HT) (N=51) | Docetaxel / Leuprolide Acetate - Deferred Treatment (D-CHT) (N=20) | Leuprolide Acetate - Deferred Treatment (D-HT) (N=17)
Hot flush (Vascular disorders) | 36 | 38 | 11 | 8
Hypertension (Vascular disorders) | 6 | 2 | 2 | 0
Flushing (Vascular disorders) | 4 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0
Venous insufficiency (Vascular disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 32 | 16 | 13 | 3
Oedema peripheral (General disorders) | 12 | 4 | 5 | 0
Asthenia (General disorders) | 5 | 3 | 5 | 1
Pyrexia (General disorders) | 5 | 2 | 0 | 0
Induration (General disorders) | 3 | 2 | 1 | 0
Mucosal inflammation (General disorders) | 4 | 0 | 1 | 0
Pain (General disorders) | 4 | 0 | 1 | 0
Chest discomfort (General disorders) | 3 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 2 | 0
Influenza like illness (General disorders) | 2 | 1 | 0 | 0
Injection site reaction (General disorders) | 3 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 1
Injection site swelling (General disorders) | 1 | 1 | 0 | 0
Localised oedema (General disorders) | 2 | 0 | 0 | 0
Tenderness (General disorders) | 2 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 1 | 0 | 0
Extravasation (General disorders) | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 0
Injection site discolouration (General disorders) | 0 | 0 | 1 | 0
Injection site discomfort (General disorders) | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0
Injection site nodule (General disorders) | 1 | 0 | 0 | 0
Injection site rash (General disorders) | 1 | 0 | 0 | 0
Necrosis (General disorders) | 0 | 0 | 1 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3 | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 4 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 16 | 4 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 2 | 6 | 0
Constipation (Gastrointestinal disorders) | 10 | 1 | 4 | 0
Stomatitis (Gastrointestinal disorders) | 7 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 3 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Buccal mucosal roughening (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 29 | 0 | 9 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 14 | 0 | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 3 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 1 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hair disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperkeratosis palmaris and plantaris (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 17 | 0 | 5 | 0
Headache (Nervous system disorders) | 14 | 3 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 2 | 3 | 0
Paraesthesia (Nervous system disorders) | 6 | 1 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 5 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 2 | 0
Ageusia (Nervous system disorders) | 2 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 2 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 2 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Sensory loss (Nervous system disorders) | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 15 | 14 | 0 | 2
Nocturia (Renal and urinary disorders) | 3 | 4 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 6 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 3 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 0
Terminal dribbling (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 15 | 17 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 2 | 2 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Genital lesion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Testicular atrophy (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 6 | 5 | 1 | 1
Depression (Psychiatric disorders) | 3 | 3 | 2 | 1
Mood altered (Psychiatric disorders) | 4 | 3 | 1 | 1
Libido decreased (Psychiatric disorders) | 2 | 4 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 1 | 0 | 0
Claustrophobia (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 4 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 2 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Anal infection (Infections and infestations) | 0 | 0 | 0 | 1
Campylobacter intestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex ophthalmic (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 6 | 8 | 3 | 2
Blood glucose increased (Investigations) | 1 | 1 | 1 | 0
Weight decreased (Investigations) | 2 | 0 | 1 | 0
Blood urea increased (Investigations) | 2 | 0 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Blood urine (Investigations) | 1 | 0 | 0 | 0
Body temperature fluctuation (Investigations) | 1 | 0 | 0 | 0
Bone density decreased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase (Investigations) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 4 | 0 | 2 | 0
Vision blurred (Eye disorders) | 4 | 0 | 0 | 0
Eye pain (Eye disorders) | 2 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 2 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Keratoconjunctivitis sicca (Eye disorders) | 1 | 0 | 0 | 0
Lacrimal disorder (Eye disorders) | 1 | 0 | 0 | 0
Optic neuropathy (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Retinopathy (Eye disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 2 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Eye penetration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 1 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Thalassaemia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study had difficulties in meeting enrollment goals within a reasonable time frame. The final sample size allowed for the safety analyses but was underpowered for drawing conclusions regarding efficacy and quality of life (QoL) endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall provide the Steering Committee a copy of any manuscript, abstract or oral communication derived from the study for review and comment at least 30 days in advance of any submission. The Sponsor's representatives shall have the right to review and/or delay any publication or presentation to prevent disclosure of Sponsor's confidential information and preserve intellectual property rights.